CLINICAL TRIAL: NCT03515772
Title: Drug-drug Interactions Between Antiretroviral Drugs and Cardiovascular Drugs in Elderly Patients From the Swiss HIV Cohort Study
Brief Title: Drug-drug Interactions Between Antiretroviral Drugs and Cardiovascular Drugs in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Thierry Buclin, Professor Dr, Centre Hospitalier Universitaire Vaudois
Other Study IDs: HIV-Interactions
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections; Drug Interactions; Cardiovascular Diseases
Keywords: dolutegravir; darunavir; amlodipine; rosuvastatin; atorvastatin
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Amlodipine with Dolutegravir: This is the "control" group regarding HIV drug interaction potential on amlodipine
- Amlodipine with Darunavir: This is the "case" group regarding HIV drug interaction potential on amlodipine
  Interventions: Drug: Co-administration of darunavir with a cardiovascular drug
- Atorvastatin with Dolutegravir: This is the "control" group regarding HIV drug interaction potential on atorvastatin
- Atorvastatin with Darunavir: This is the "case" group regarding HIV drug interaction potential on atorvastatin
  Interventions: Drug: Co-administration of darunavir with a cardiovascular drug
- Rosuvastatin with Dolutegravir: This is the "control" group regarding HIV drug interaction potential on rosuvastatin
- Rosuvastatin with Darunavir: This is the "case" group regarding HIV drug interaction potential on rosuvastatin
  Interventions: Drug: Co-administration of darunavir with a cardiovascular drug

INTERVENTIONS:
Drug: Co-administration of darunavir with a cardiovascular drug — Co-administration of darunavir, an HIV agent considered prone to induce drug interactions, with a cardiovascular drug (amlodipine, atorvastatin or rosuvastatin). Note that a patient will be able to participate in the intervention group and the control group if a change in his/her anti-HIV treatment occurs (study partly parallel and partly in cross-over).
  Groups: Amlodipine with Darunavir; Atorvastatin with Darunavir; Rosuvastatin with Darunavir

SUMMARY:
Ageing is characterized by physiological changes, which can impact drug pharmacokinetics and thereby cause drug-drug interactions. This study aims to assess the pharmacokinetics of amlodipine, atorvastatin and rosuvastatin in the presence of darunavir/ritonavir (inhibitor of drug metabolizing enzymes and drug transporters), by comparison with dolutegravir (no inhibitory effects on cytochromes or transporters involved in the disposition of the evaluated co-medications), in order to characterize the importance of drug-drug interactions in elderly individuals.

DETAILED DESCRIPTION:
HIV-infected individuals live longer, making the proportion of older individuals within the HIV infected population constantly growing. Thus, the management of HIV infection is becoming more complex as patients encounter more age related chronic ailments such as hypertension, diabètes and tumors, or acute diseases, sometimes severe, leading to polypharmacy and consequently to potential drug-drug interactions (DDI). In addition, aging is characterized by a decline in the function of elimination organs, which may impact the pharmacokinetics of drugs and thereby the magnitude of DDI.

The principal aim of the study is to determine the importance of DDIs between antiretroviral drugs and commonly prescribed co-medications (namely amlodipine, rosuvastatin and atorvastatin) in HIV-infected patients of the Swiss HIV Cohort Study (SHCS). The investigation will include a majority of patients over 60 years old, yet without excluding younger patients. Pharmacokinetic investigations will be primarily conducted in patients treated with darunavir/ritonavir- or dolutegravir-containing regimens, and who receive one of the cardiovascular drug of interest. The objective is to contrast the effects of darunavir/ritonavir (strong inhibitor of drug metabolizing cytochromes) and dolutegravir (devoid of inhibitory effects on these enzymes), in order to determine the magnitude of the interaction with the co-medication. Besides their common use in elderly HIV-infected patients, amlodipine, atorvastatin and rosuvastatin were primarily selected due to their predisposition to become victims of drug-drug interactions. In addition, the same study framework will possibly serve to examine further drug combinations susceptible to interact, whose exploration could be of interest from a clinical point a view to stimulate future confirmatory research. It will thus be open to investigate associations of other cardiovascular agents with the antiretroviral drugs defined above, or with other antiretroviral drugs.

On a morning selected for investigation, the patient will take the antiretroviral medications together with the comedication of interest with a standard breakfast. Serial blood samples will be collected into EDTA-K monovettes (2.7 ml) from a catheter positioned in the forearm at the following time-points: t = 0 (just before the drug intake) and 30 minutes, 1, 2, 3, 4, 6, 8, 10, and 12 hours after drug intake (a certain flexibility in sampling times is allowed, provided that dosing and sampling times are carefully recorded). The patient will then spend the night at home and return the following morning to provide the last sample of blood 24 hours after drugs intake. In total, 30 ml of blood will be required for a full pharmacokinetic investigation).

A second full pharmacokinetic investigation will be performed for patients undergoing antiretroviral treatment change for clinical reasons. The investigation will be scheduled two weeks after switching treatment, so that a steady-state is reached, and will be performed as described above.

The blood samples will be centrifuged and the separated plasma will be frozen at -80°C until analysis by liquid chromatography tandem mass spectrometry (LC-MS/MS). Pharmacokinetic parameters will be first estimated by classical non-compartmental approaches: Maximal concentration (Cmax), minimal concentration (Cmin), Area Under the Curve (AUC), slope of the terminal phase (Lambda_z), clearance (Cl), half-life (t1/2). These parameters will be compared according to the co-prescription of darunavir/ritonavir versus dolutegravir, using a variance analysis on log-transformed values. The analysis will accommodate partial pairing of parameter values obtained in patients investigated in cross-over, through the inclusion of a random patient factor (assumed to take independent values only between patients). PK parameters of antiretroviral drugs will be simply described.

ELIGIBILITY:
Inclusion Criteria:

* documented HIV-infection
* informed consent as documented by signature (Appendix Informed Consent Form)
* included in the SHCS and followed-up in the HIV Clinic in Lausanne or in Basel
* treatment with a HIV therapy including either once-daily ritonavir-boosted darunavir or dolutegravir (or others ARV drugs for the exploratory investigations)
* treatment with one or eventually 2 of the comedications of interest, i.e. amlodipine, atorvastatin or rosuvastatin (or any drug potentially involved in clinically relevant DDI for the exploratory investigations).
* Ability to comply with the study requirements

Exclusion Criteria:

* Presence of severe comorbidities (i.e. cirrhosis (Child-Pugh score C), heart failure (NYHA 3-4), advanced kidney impairment (KDOQI 4-5)) which can substantially impact the pharmacokinetic of drugs and significantly confound the study results.
* Presence of interacting non HIV comedications (i.e comedications with known, strong inhibitory or inducing effects on drug metabolizing cytochromes and drug transporters, which might significantly confound the study results)
* Participants incapable of jugement or participants under tutelage
* Known or suspected non-compliance, drug or alcohol abuse considered at risk to significantly confound the study results
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia of the participant,
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Women who are pregnant or breastfeeding

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: HIV patients treated with the anti-HIV agents dolutegravir or darunavir, while simultaneously receiving cardiovascular agents, namely amlodipine, atorvastatin or rosuvastatin
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Circulating exposure (AUC) to cardiovascular agent amlodipine | 2 weeks
  Area under the curve (AUC) of the cardiovascular drug, namely amlodipine, in the presence of darunavir/ritonavir (inhibitory effect hypothesized) or dolutegravir (no inhibitory effect predicted).
Circulating exposure (AUC) to cardiovascular agent atorvastatin | 2 weeks
  Area under the curve (AUC) of the cardiovascular drug, namely atorvastatin in the presence of darunavir/ritonavir (inhibitory effect hypothesized) or dolutegravir (no inhibitory effect predicted).
Circulating exposure (AUC) to cardiovascular agent rosuvastatin | 2 weeks
  Area under the curve (AUC) of the cardiovascular drug, namely rosuvastatin in the presence of darunavir/ritonavir (inhibitory effect hypothesized) or dolutegravir (no inhibitory effect predicted).

SECONDARY OUTCOMES:
Circulating exposure (AUC) to another cardiovascular agent, if one appears frequently associated with HIV agents | 2 weeks
  Area under the curve (AUC) of the cardiovascular drug in the presence of darunavir/ritonavir (inhibitory effect hypothesized) or dolutegravir (no inhibitory effect predicted).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Buclin, Prof., Principal Investigator — Service of Clinical Pharmacology
Locations (2):
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share anonymized IPD with colleagues interested upon motivated request
Supporting Information: Study Protocol, ICF
Time Frame: after end of study and publication
Access Criteria: Motivated request

REFERENCES:
- [Derived] Courlet P, Guidi M, Alves Saldanha S, Stader F, Traytel A, Cavassini M, Stoeckle M, Buclin T, Marzolini C, Decosterd LA, Csajka C; and the Swiss HIV Cohort Study. Pharmacokinetic/Pharmacodynamic Modelling to Describe the Cholesterol Lowering Effect of Rosuvastatin in People Living with HIV. Clin Pharmacokinet. 2021 Mar;60(3):379-390. doi: 10.1007/s40262-020-00946-3. Epub 2020 Oct 29. PMID 33124006
- See also: Website of the Service of Clinical Pharmacology at CHUV, Lausanne — http://www.chuv.ch/fr/pcl/